CLINICAL TRIAL: NCT06165484
Title: Evaluation of Patients of Failed in Vitro Fertilization Cycle: Prospective Cohort Study
Brief Title: Laparoscopy in Failed IVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Saber Ali, Assistant Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: failed IVF
Record Dates: First submitted 2023-11-20; First posted 2023-12-11 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Laparoscopy; Hysteroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with failed ivf cycle (Experimental)
  Interventions: Procedure: laparoscopy and hysteroscopy

INTERVENTIONS:
Procedure: laparoscopy and hysteroscopy — laparoscopy and hysteroscopy for patient with failed IVF

SUMMARY:
Current in-vitro fertilization (IVF) consumers are enjoying better success rates than early seekers, but only about a quarter of IVF cycles result in a live birth and many patients remain infertile after multiple IVF attempts. Recurrent IVF failure is distressing to patients and challenging to clinicians. Despite interventions have been proposed to improve IVF outcome after couples of failed cycles, only a few of which are evidence based.

Laparoscopy, as the gold standard for the evaluation of the pelvis, was used to be the routine procedure for many reproductive physicians. It provides information on endometriosis, tubal patency, and pelvic adhesions and a chance to fix these lesions concurrently.

DETAILED DESCRIPTION:
Current in-vitro fertilization (IVF) consumers are enjoying better success rates than early seekers, but only about a quarter of IVF cycles result in a live birth and many patients remain infertile after multiple IVF attempts. Recurrent IVF failure is distressing to patients and challenging to clinicians. Despite interventions have been proposed to improve IVF outcome after couples of failed cycles, only a few of which are evidence based.

Laparoscopy, as the gold standard for the evaluation of the pelvis, was used to be the routine procedure for many reproductive physicians. It provides information on endometriosis, tubal patency, and pelvic adhesions and a chance to fix these lesions concurrently.

The role of laparoscopy, especially in women whose normal screening tests suggest that pelvic pathology seem to be unlikely. However, sometimes a "normal" pelvic imaging can be misleading, since HSG or ultrasonography cannot to rule out hydrosalpinx and endometriosis completely. Furthermore, it has been shown that HSG is insufficient for predicting tubal potency for some patients with risk of pelvic adhesions, with a sensitivity between 0.0% and83% and specificity between 50% and 90%. When initial IVF treatments fail, can we offer the couples to choose additional cycle of IVF instead of evaluation of the potential peritoneal factor? In cases of otherwise so called "Unexplained infertility", the investigation cannot be considered complete until laparoscopy has been performed.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patients ages ranged from 20 to 40 years. 2. menstrual cycles with a duration of 24 to 38 days and no ovulatory dysfunction. 3. normal findings of pelvic ultrasonography and HSG assessment, without visible lesions that could cause implantation failure, for example: endometrial polyps, submucosal myomas, uterine septum and intrauterine adhesions.

  4. hormonal values were within the normal range. 5. Semen analyses were normal according to the World Health Organization (WHO) 2010 criteria.

  6. no previous surgical treatment for endometriosis; no previous oophorectomy or salpingectomy.

  7. Patients included in the study had failed to conceive after at least one cycles of IVF-ET when indicated.

Exclusion Criteria:

- 1. Couples with severe male factor infertility. 2. Premature ovarian failure. 3. Patients with a poor ovarian reserve and poor responders. 4. Contraindication to laparoscopy such as mechanical or large abdominal mass (> 24 weeks gestation size).

5. Contraindication to hysteroscopy such as recent or active pelvic inflammatory disease and active uterine bleeding.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Improving the pregnancy outcome in patients with recurrent IVF failure. | 1.5 YEARS
  To assess if the diagnosis and treatment of pelvic or uterine pathologies with laparoscopy and hysteroscopy is of role in improving the pregnancy outcome (live birth rate and ongoing pregnancy rate) in patients with recurrent IVF failure .

SECONDARY OUTCOMES:
Abnormal laparoscopy findings and surgery-related complications | 1.5 YEARS

IPD SHARING:
Plan to Share IPD: Undecided